CLINICAL TRIAL: NCT07193329
Title: Psychological Distress in Malignant Tumor Patients: Effects on Treatment Adherence, Outcomes, and Quality of Life
Status: Recruiting | Type: Observational
Sponsor: Gang Chen, MD (Other)
Responsible Party: Sponsor-Investigator, Gang Chen, MD, M.D., Ph.D., Professor, First Affiliated Hospital of Wenzhou Medical University
Organization: First Affiliated Hospital of Wenzhou Medical University (Other)
Other Study IDs: KY2025-235
Record Dates: First submitted 2025-07-22; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Psychological Distress; Malignant Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Malignant Tumor Patients with Psychological Distress
- Malignant Tumor Patients without Psychological Distress

SUMMARY:
The goal of this observational study is to learn about the Psychological Distress in Malignant Tumor Patients about Effects on Treatment Adherence, Outcomes, and Quality of Life. The main question it aims to answer is:

Does Psychological Distress affect Malignant Tumor Patients' Effects on Treatment Adherence, Outcomes, and Quality of Life? Malignant Tumor Patients with or without Psychological Distress will answer GAD-7 and PHQ-9 and their Treatment Adherence, Outcomes, and Quality of Life be recorded for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* (1) Confirmed malignant tumors by imaging or pathology (such as hepatobiliary carcinoma, gastric cancer, breast cancer, lung cancer, etc.)
* (2) Planning to receive or currently undergoing systemic treatment (such as surgery, chemotherapy, TACE, targeted therapy, etc.)
* (3) Age ≥18 years old
* (4) Sign the informed consent form and voluntarily participate in this study

Exclusion Criteria:

* (1) Combined with severe systemic diseases (such as severe cardiovascular and cerebrovascular diseases)
* (2) There is severe cognitive impairment and it is impossible to complete the questionnaire assessment
* (3) Incomplete clinical data or loss to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malignant tumors who were treated at the First Affiliated Hospital of Wenzhou Medical University from July 2025 to July 2028
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by mRECIST (%) | at 4-12 weeks after treatment initiation.
  Proportion of participants achieving complete response (CR) or partial response (PR) based on mRECIST criteria, measured on contrast-enhanced CT/MRI.

OTHER OUTCOMES:
PFS(months) | through study completion, an average of 3 years
  PFS defined as time from treatment initiation to radiologically confirmed disease progression (mRECIST) or death from any cause, whichever occurs first.
Quality of Life (EORTC QLQ-C30) | through out treatment, average of 3 years
  Quality of life will be assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30), with change from baseline analyzed at follow-up intervals.
Treatment Adherence (MMAS-8) | within one month after treatment
  Adherence will be evaluated by researchers using the 8-item Morisky Medication Adherence Scale (MMAS-8).
OS (month) | through study completion, an average of 3 years
  OS defined as time from treatment initiation to death from any cause.
PHQ-9 | baseline
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item self-report tool designed to screen for and assess the severity of depressive symptoms based on DSM criteria.
GAD-7 | baseline
  The Generalized Anxiety Disorder-7 (GAD-7) is a 7-item questionnaire used to identify and grade the severity of generalized anxiety symptoms.
HAMD | baseline
  The Hamilton Depression Rating Scale (HAMD) is a clinician-administered instrument widely used to evaluate the severity of depressive disorders in clinical and research settings.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected throughout the trial
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The individual participant data (IPD) that underlie the results reported in this article will be made available beginning 6 months after publication and ending 36 months after publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal for use in achieving the aims of a specified research project. Proposals should be directed to corresponding author's email. To gain access, data requesters will need to sign a data access agreement.